CLINICAL TRIAL: NCT01346059
Title: Intracolonic Vancomycin Therapy in Severe C. Diff Colitis: A Double Blinded Randomized Prospective Trial
Brief Title: Intracolonic Vancomycin Therapy in Severe C. Diff Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues with catheter placement; researcher left institution
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-195
Record Dates: First submitted 2011-03-03; First posted 2011-05-02 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2016-12

CONDITIONS: Colitis
Keywords: Clostridium; Colitis; Intracolonic vancomycin; psuedomembranous colitis
MeSH Terms: conditions — Colitis | interventions — Vancomycin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator): The saline arm will receive normal saline through the catheter as a placebo.
  Interventions: Drug: Saline
- Vancomycin (Experimental): The vancomycin arm will receive vancomycin solution through the catheter.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Vancomycin solution will be instilled through the colonic catheter every 6 hours. 250cc of solution will be used each time. The solution is 2 grams vancomycin mixed in 1 liter normal saline.
  Other Names: Vancocin
  Arms: Vancomycin
Drug: Saline — Saline, used as a placebo, will be instilled through the colonic catheter. Every 6 hours, 250cc of saline will be used.
  Other Names: Normal Saline
  Arms: Saline

SUMMARY:
Clostridium difficile is a bacteria that can infect the colon and cause severe diarrhea in patients after recent antibiotic use. The current standard of care treatment for severe C. diff. consists of oral vancomycin and/or intravenous metronidazole. When treatment is unsuccessful, it can lead to need for removal of the entire colon or even death. In fact, mortality rates in the literature range from 11-37% for C. diff. The most commonly quoted mortality rate is 14% for severe infection. It is believed that the failure of treatment may stem from an adynamic ileus (paralysis of the small bowel). This ileus may prevent the oral vancomycin from reaching the colon and therefore it does not treat the problem. Vancomycin functions by direct contact with the colon. Therefore, if the vancomycin is instilled directly into the colon, it can come into contact with and be its intended target. : The objective of the study is to improve treatment of severe C. diff. colitis . C. diff. infection is defined as severe if there is evidence of ileus accompanied by any one of the following: fever greater than 38.30C, , acidemia, serum albumin less than 2.5, or white blood cell count greater than 14,000.

DETAILED DESCRIPTION:
Patients in the surgical intensive care unit with severe C. diff. are eligible and if consented will be randomized in a 1:1 ratio to a control group or the treatment group. Each group will undergo a colonoscopy on day one of the study. A 14 French Cook colonic decompression catheter will be placed at that time. This catheter is a 175cm long soft flexible catheter designed to be placed in the colon. Its usual use is to remove air from a colon that is dilated. The catheter is placed into the colon by first placing a guidewire through the colonoscope. The colonoscope is then removed leaving the guidewire in place. The catheter is then thread into the colon over the guidewire. An xray is obtained to confirm the location of the catheter and then the guidewire is removed. The guidewire is a very thin, soft, flexible wire. The patient will not have any undue discomfort secondary to the catheter. The control group will have 250cc of sterile saline solution instilled through the catheter into the colon every 6 hours. The study group will have 250cc of vancomycin solution instilled every 6 hours. The solution will be 2 grams vancomycin dissolved in a 1 liter normal saline irrigation bottle. The catheter will be clamped in both groups after instillation until the next treatment. Of note, both groups will receive the current standard treatment of 500mg IV metronidazole every 8 hours and 250mg oral vancomycin every 6 hours throughout the study. Every day the patients will have a blood draw to check the white blood cell count as is the current practice. The patients will also have a vancomycin trough level checked via blood test. This will occur just prior to the first dosing on treatment day number 3. This will be a blinded lab value as to not unblind the investigators. At resolution Patients will undergo a repeat colonoscopy when there is a decrease of diarrhea (less than 3 stools daily) and a normalized white blood cell count or on day 7 if symptoms persist. The expected length of treatment is approximately 7 days. If there is no improvement at fourteen days, the trial will be stopped for futility. The trial will also be halted if the attending physician determines that the patient needs surgery or if the clinical status of the patient has deteriorated to a point where keeping the patient enrolled will potentially cause harm. Follow-up after completing the trial will consist of phone interviews to screen for recurrence of infection. A weekly phone call will be made for the first three weeks and then two monthly calls will take place after that for a total of three months follow-up. The primary investigator will make these phone calls.

ELIGIBILITY:
Inclusion Criteria:

* SICU patient
* positive c. diff toxin assay
* visualization of pseudomembranes on colonoscopy,
* able to give consent or have representative to give consent.

Exclusion Criteria:

* Under age 18
* pregnant
* absence of a colon or surgical discontinuity of bowel
* allergy to vancomycin
* need for anti-diarrheal medication
* need for prolonged antibiotics for other cause
* need for probiotics
* need for other medications with action against C. diff.
* need for surgery, colon perforation
* recent IV IG use
* toxic megacolon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc B Grodsky, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients enrolled undergo a complete colonoscopy with placement of a 14 French colon decompression catheter (Cook Medical). Proper placement of the catheter in the cecum is verified by abdominal X-ray. Patients are randomized to either Saline or Vancomycin arms.
Period: Overall Study
Arm/Group | Saline | Vancomycin
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Vancomycin | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Diarrhea and White Blood Cell Count Elevation
Description: If the patient has resolution of diarrhea, white blood cell count, and abdominal pain, the protocol will be stopped.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Vancomycin
Number analyzed (Participants) | 0 | 1
Participants |  | 1

2. Secondary Outcome: Mortality
Description: Death within 30 days of enrollment, in or out of hospital
Time Frame: 30 day
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Vancomycin
Number analyzed (Participants) | 0 | 1
Participants |  | 0

3. Secondary Outcome: Need for Colectomy
Description: Partial or complete colectomy performed within 30 days of enrollment
Time Frame: 30 day
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Vancomycin
Number analyzed (Participants) | 0 | 1
Participants |  | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Saline | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Technical problems with catheters becoming dislodged from the ideal site of placement (cecum) leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No